CLINICAL TRIAL: NCT05232591
Title: Evaluation of IL-17, TNF-alpha, RANKL Levels in Gingival Cervicular Fluid of Teeth With Periapical Lesions Diagnosed With Chronic Apical Periodontitis
Brief Title: Evaluation of IL-17, TNF-alpha, RANKL Levels in Gingival Cervicular Fluid
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Esin Özlek, Asist. Prof., Yuzuncu Yil University
Other Study IDs: 2021/08-02
Record Dates: First submitted 2022-01-17; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Apical Periodontitis
Keywords: Gingival cervicular fluid; IL-17; TNF-alpha; RANKL
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The gingival cervicular fluid is a biological fluid originating from blood plasma, present in different compositions in the gingival sulcus, and has the characteristics of exudate, which determines the ecology of the gingival sulcus. Cellular components (epithelium, bacteria, leukocytes, erythrocytes, leukocytes, viruses and their by-products), electrolytes, bacterial-metabolic products, cytokines, host and bacterial enzymes and enzyme products-inhibitors (acid phosphatase, alkaline phosphatase, aspartate aminotransferase, lactate dehydrogenase, aryl sulfatase, etc.), and immunoglobulins form the characteristic features of the fluid, revealing the importance of this fluid in terms of periodontal disease.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: GCF samples will be taken from the teeth diagnosed with chronic apical periodontitis
  Interventions: Diagnostic Test: The teeth diagnosed with chronic apical periodontitis
- 2: GCF samples will be taken from the collateral teeth (healthy teeth) of the teeth diagnosed with chronic apical periodontitis.
  Interventions: Diagnostic Test: The teeth diagnosed with chronic apical periodontitis

INTERVENTIONS:
Diagnostic Test: The teeth diagnosed with chronic apical periodontitis — GCF samples will be taken from the teeth diagnosed with chronic apical periodontitis

SUMMARY:
Inflammatory process begins around root apex as a result of bacterial infection of pulp cavity in chronic apical periodontitis. Bone destruction can begin in apical region after immunological reactions at the end of inflammatory process, and radiolucent periapical lesion seems in this way. If bone destruction around apical region is in the rate of 30%, we can notice this difference eventually. Histological manifestations of periapical inflammation can be observed in the result of pulp necrosis and inflammation around apical region. Mocelular methods can determine the type of therapy in various diseases. Each region and tissue reserve specific host factors. Vast majority of pulpal inflammation was trigerred by microorganisms. Certain bacterial virulence factors may damage host tissue directly, other virulence factors can stimulate prolonged non-specific immune response causing tissue damage. In the last phase of infection, immunopathological destruction of pulp tissue is observed due to humoral response. IL-17 is an important inflammatory cytokine released from T cells of the immune system. TNF-alpha and RANKL are also mediators responsible for bone destruction metabolism. TNF is a cytokine mediating immunologic changes during periodontal disease. TNF induction stimulate secondary mediators taking part as chemotactic cytokines. TNF has two different types; TNF-alpha and TNF-beta. TNF-alpha is a polypeptide cytokine produced by macrophages and monocytes. TNF-alpha stimulates bone resorption . There has been limited researches analyzing GCF, blood and tissue of pulp, dentin-derived fluid and periapical fluid for molecular diagnosis so far. GCF is a fluid derived from gingival groove. This fluid contains a lot of host factors such as anticor, bacterial antigen, protein and cytokines. GCF sampling is a non-invasive method, it can be used to provide diagnostic information in all clinical cases. In this study, we will evaluate the levels of IL-17, TNF-alpha and RANKL in the gingival crevicular fluid of teeth with periapical lesion diagnosed with chronic apical periodontitis. Thus, it will be evaluated whether these markers can be used for diagnosis and follow-up of the disease in teeth with periapical lesions.

DETAILED DESCRIPTION:
It is planned to include volunteer patients who came to Van YYU Faculty of Dentistry, Oral and Maxillofacial Radiology Department between February and March 2022 for routine examination. Patients who applied to Yüzüncü Yıl University Faculty of Dentistry for treatment and met the study criteria will be included in the study by signing an informed consent form. 40 patients diagnosed with chronic apical periodontitis and having teeth with radiographic periapical lesions will be included in the study. Patients with periodontitis will not be included in the study.

GCF samples will be taken from the teeth diagnosed with chronic apical periodontitis and the contralateral teeth (from healthy teeth). The tooth which is resource of GCF will be isolated with cotton pellets. After the supragingival plaque is carefully removed with a curette, the tooth will be air-dried for 10 seconds, and periopaper strips will be placed in the gingival sulcus until resistance is felt. Periopaper strips will be removed from the gilgival sulcus after 1 minute. The levels of IL-17, TNF-alpha and RANKL from the samples in the gingival crevicular fluid will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons between the ages of 18 and 45 years
* Mandibular molar teeth that were diagnosed with symptomatic irreversible pulpitis and periapical lesion

Exclusion Criteria:

* Patients who are taken analgesic inflammatory drugs with in the last 12 hours
* Pregnancy or lactation
* Teeth with periodontal diseases
* Teeth with sensitive to percussion and palpation
* Teeth with root resorption
* Teeth with immature/open apex

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: It is planned to include volunteer patients who came to Van YYU Faculty of Dentistry, Oral and Maxillofacial Radiology Department for routine examination.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
IL-17 Level | 6 months
  Concentration of IL-17 in GCF
TNF-alpha | 6 months
  Concentration of TNF-alpha in GCF
RANKL | 6 months
  Concentration of RANKL in GCF

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Newton CW, Hoen MM, Goodis HE, Johnson BR, McClanahan SB. Identify and determine the metrics, hierarchy, and predictive value of all the parameters and/or methods used during endodontic diagnosis. J Endod. 2009 Dec;35(12):1635-44. doi: 10.1016/j.joen.2009.09.033. PMID 19932338
- [Result] Ricucci D, Siqueira JF Jr, Bate AL, Pitt Ford TR. Histologic investigation of root canal-treated teeth with apical periodontitis: a retrospective study from twenty-four patients. J Endod. 2009 Apr;35(4):493-502. doi: 10.1016/j.joen.2008.12.014. PMID 19345793